CLINICAL TRIAL: NCT01778790
Title: Assessment of Efficacy, Safety and Effects on Quality of Life of Deep Brain Stimulation to the Medial Forebrain Bundle in Patients With Treatment Resistant Major Depression (FORESEE II: FOREbrain Stimulation dEprEssion)
Brief Title: Deep Brain Stimulation of the Superolateral Branch of the Medial Forebrain Bundle (slMFB) for the Treatment of Refractory Major Depression
Acronym: FORESEEII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Thomas E. Schlaepfer, MD, Professor of Psychiatry and Psychotherapy, University Hospital, Bonn
Masking: Double | Purpose: Treatment
Other Study IDs: BSG-13-2319DBS
Record Dates: First submitted 2013-01-18; First posted 2013-01-29 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Deep Brain Stimulation
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham Stimulation for 8 weeks (Sham Comparator): Implantation of internal pulse generator (IPG), Sham Stimulation
  Interventions: Device: Deep Brain Stimulation with Activa PC Multi-program Neurostimulator
- Stimulation for 8 weeks (Active Comparator): Implantation of IPG and active stimulation
  Interventions: Device: Deep Brain Stimulation with Activa PC Multi-program Neurostimulator

INTERVENTIONS:
Device: Deep Brain Stimulation with Activa PC Multi-program Neurostimulator — Device: DBS 130 Hertz (Hz) frequency, 90us pulsewidth, 4 Volt (V) currency Amplitude
  Device: DBS - No Stimulation (Sham) 130 Hertz (Hz)frequency, 90us pulsewidth, 0 Volt (V) currency Amplitude

SUMMARY:
The investigators will investigate in a sham controlled staggered onset design antidepressant effects and safety of deep brain stimulation (DBS) to the superolateral branch of the main medial forebrain bundle (slMFB).

DETAILED DESCRIPTION:
The target point for DBS in major depression disorder is located lateral to the ventral tegmental area (VTA) in the midbrain at the branching point of the superolateral branch (slMFB) from the main medial forebrain bundle (MFB).

The exact stimulation coordinates are:

Montreal Neurologic Institute brain 152 coordinates (MNI152 coordinates):

left: x(lat.)=-5, y(ap)=-14, z(vert.)=-8 right: x(lat.)=5, y(ap)=-14, z(vert.)=-9

Mid-commissural point coordinates (MCP coordinates):

eft: x(lat.)=-6, y(ap)=-1, z(vert.)=-6 right: x(lat.)=4, y(ap)=-1, z(vert.)=-7

All coordinates refer to the MNI152 brain.

Legend:

slMFB = superolateral branch of medial forebrain bundle lat. = lateral, ap= anteroposterior, vert. = vertical.

More information can be found at: http://goo.gl/n9sWV

ELIGIBILITY:
Inclusion Criteria:

* Major depression (MD), severe, unipolar
* German mother tongue
* Age 20 to 75 Years
* Hamilton Depression Rating Scale (HRSD24) score of > 21
* Global Assessment of Function (GAF) score of < 45
* At least 4 episodes of depression or chronic episode > 2 years
* Failure to respond to

  * adequate trials (>5 weeks at the maximum recommended or tolerated dose) of primary antidepressants from at least 3 different classes;
  * adequate trials (>3 weeks at the usually recommended or maximum tolerated dose) of augmentation/combination of a primary antidepressant using at least 2 different augmenting/combination agents (lithium, T3, stimulants, neuroleptics, anticonvulsants, buspirone, or a second primary antidepressant);
  * an adequate trial of electroconvulsive therapy (ECT) (>6 bilateral treatments) and; an adequate trial of individual psychotherapy (>20 sessions with an experienced psychotherapist)
* Able to give written informed consent
* Compliance to participate in the study
* Drug free or on stable drug regimen at least 6 weeks before study entry

Exclusion Criteria:

* Current or past non-affective psychotic disorder
* Any current clinically significant neurological disorder or medical illness affecting brain function, other than motor tics or Gilles de la Tourette syndrome
* Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI)
* Any surgical contraindications to undergoing DBS
* Current or unstably remitted substance abuse (aside from nicotine)
* Pregnancy and women of childbearing age not using effective contraception
* History of severe personality disorder
* Acute suicidal tendency

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Depression Severity assessed with Montgomery Asberg Depression Scale (MADRS) | 6 and 12 month after DBS stimulation onset
  Change in MADRS after 6 and 12 months as compared to mean baseline score and one month placebo treatment. MADRS is a ten-item diagnostic questionnaire which psychiatrists use to measure the severity of depressive episodes in patients with mood disorders. It is used as an adjunct to the Hamilton Rating Scale for Depression (HAMD) and more sensitive to the changes in depression than the Hamilton Scale is.

SECONDARY OUTCOMES:
Depression Severity rated with Hamilton Depression Rating Scale (HDRS24) | 6 and 12 month after DBS stimulation onset
  The Hamilton Rating Scale for Depression (HRSD), also known as the Hamilton Depression Rating Scale (HDRS) or abbreviated to HAM-D, is a multiple choice questionnaire that clinicians may use to rate the severity of a patient's major depression. The questionnaire rates the severity of symptoms observed in depression such as low mood, insomnia, agitation, anxiety and weight loss. The questionnaire is presently one of the most commonly used scales for rating depression in medical research.
  Measures will be taken at same time points as primary outcome measure.

OTHER OUTCOMES:
Comprehensive neuropsychological test battery | 6 and 12 month after DBS stimulation onset
Adverse Event Schedule | 6 and 12 month after DBS stimulation onset
  Adverse events will be recorded during the study using a structured questionnaire. All possible adverse events (AEs) are assessed in severity, duration and actions taken. 12 months after stimulation onset results will be compiled and rated as being due to the surgical procedure, device, or stimulation. Serious adverse events (SAEs) will be discussed individually if a modification of study protocol is required.
  Additional, there will be a safety and efficacy analysis after 6 implanted patients.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E. Schlaepfer, MD, Principal Investigator — University Hospital, Bonn; Volker Coenen, MD, Principal Investigator — University Hospital Freiburg
Locations (1):
- University Hospital Bonn, Bonn, Germany

REFERENCES:
- [Derived] Kilian HM, Meyer DM, Bewernick BH, Spanier S, Coenen VA, Schlaepfer TE. Discontinuation of Superolateral Medial Forebrain Bundle Deep Brain Stimulation for Treatment-Resistant Depression Leads to Critical Relapse. Biol Psychiatry. 2019 Mar 15;85(6):e23-e24. doi: 10.1016/j.biopsych.2018.07.025. Epub 2018 Sep 22. No abstract available. PMID 30253883
- See also: DBS target site description — http://tiny.cc/sl-mfb